CLINICAL TRIAL: NCT04213066
Title: Stochastic Resonance Applied to Amblyopia Training and the Plasticity of Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-BR-102-050-t
Record Dates: First submitted 2019-12-22; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Amblyopia; Amblyopia, Anisometropic
Keywords: Amblyopia; Amblyopic training; Contrast sensitivity; Grating acuity; Stochastic resonance; Visual acuity; Visual evoked potential
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): This group received eye-hand practice for drawing pictures.
  Interventions: Device: Portable tablet
- Grating group (Experimental): This group received eye-hand practice for drawing pictures with rotating grating stimuli of various spatial frequencies.
  Interventions: Device: Portable tablet
- Random dot group (Experimental): This group received eye-hand practice for drawing pictures with rotating grating stimuli of various spatial frequencies constructed by random dots of stochastic resonance.
  Interventions: Device: Portable tablet

INTERVENTIONS:
Device: Portable tablet — Each training session was limited to 15 minutes a day, 5 days a week. The entire training period was 6 months.

SUMMARY:
The prevalence of Taiwan's population with amblyopia is 2-5%. Amblyopia affects the daily life and learning ability. The human visual system can be developed normally with exposure of clear images on the retina, which often drive the development and projection of optic nerves progressively. In general, the visual acuity progresses gradually with age. A normal vision is relatively mature until 8 years old. Several types of amblyopia (strabismic amblyopia, refractive amblyopia, and deprivation amblyopia) are identified. The refractive amblyopia and deprivation amblyopia must be corrected by wearing glasses or surgeries. Otherwise, amblyopia is often corrected by occlusion of the dominant eye or amblyopia training. The Cambridge Stimulator (CAM) with rotating grating is commonly used in clinic in Taiwan. The principle of the CAM allows subjects to draw pictures on the plate in coincidence with occlusion of the dominant eye. The parents have to go with their children to a hospital weekly. The CAM training is a stereotyped visuomotor behavior, which usually causes fatigue and uninteresting results for children.

Recently, some computer games have been incorporated with CAM training. However, their clinical impact on amblyopia is largely unknown. Moreover, most of studies don't have long-term tracking, and they only use limited assessments. In this project, a home-based training would be built for children with amblyopia. A CAM training with a hierarchical structure with story-based organization would be implemented in the tablet. It will save time for children and parents for traffic between the home and hospital. The CAM training with organized structure would increase acceptability and create subjects' motivation for long-term training. In addition, a stochastic resonance theory would be incorporated with the CAM training to potentiate the learning curve of a visuomotor skill in young children. Five systematic assessments, including visual acuity, grating acuity, contrast sensitivity, and 2 measurements of visual evoked potentials (VEPs), would be used. The investigators hypothesized that the rotating grating stimulation and stochastic resonance stimulation groups showed significant enhancement of the visual functions compared with the control group and performance of the VEPs toward better eye through the home-based training apparatus.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were 4-8 years old.
2. Participant had binocular or monocular best-corrected visual acuity (BCVA) of ≤0.8, or they exhibited binocular BCVA difference of ≥0.2.
3. Participant had the wearing of optimal spectacle correction.

Exclusion Criteria:

1. Children with deprivation amblyopia were excluded.
2. Children with ptosis were excluded.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Visual acuity (VA) | Change from Baseline VA at 1, 2, 3 and 6 months
  Landolt C chart was used.
Grating acuity (GA) | Change from Baseline GA at 1, 2, 3 and 6 months
  Horizontal or vertical square-wave grating stimuli were used.
Contrast sensitivity (CS) | Change from Baseline CS at 1, 2, 3 and 6 months
  Circular-shape horizontal square-wave grating stimuli were used.
Visual evoked potential (VEP) | Change from Baseline VEP at 1, 2, 3 and 6 months
  Transient VEP and Steady state VEP of the Cortical EEG were recorded.

SECONDARY OUTCOMES:
Total practice duration | Throughout 6 months
  Practice duration was recorded in the tablet.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Zen Shaw, Professor, Principal Investigator — Department of Pyschology, National Cheng Kung University

REFERENCES:
- [Derived] Yeh WH, Lai LJ, Chang DW, Lin WS, Lin GM, Shaw FZ. Portable rotating grating stimulation for anisometropic amblyopia with 6 months training. Sci Rep. 2021 Jun 1;11(1):11430. doi: 10.1038/s41598-021-90936-7. PMID 34075118